CLINICAL TRIAL: NCT02099773
Title: Support Staff's Interactions With Adults With Intellectual Disability Who Use Augmentative and Alternative Communication
Brief Title: Support Staff-client Interactions With Augmentative and Alternative Communication
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S56517
Record Dates: First submitted 2014-03-24; First posted 2014-03-31 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-11

CONDITIONS: Intellectual Disability
Keywords: AAC; support worker; direct care staff; intellectual disability; learning disability; communication; adults
MeSH Terms: conditions — Intellectual Disability; Learning Disabilities; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- support workers & AAC users: Support workers who use KeyWordSigning in the communication with their client who has an intellectual disability
- support workers & KWS users: Support workers who use aided AAC in the communication with their client who has an intellectual disability

SUMMARY:
This exploratory and observational study focuses on adults with an intellectual disability (ID) and their support workers. Two groups of clients are observed: clients using Key Word Signing, and clients using aided Augmentative and Alternative Communication (AAC). Approximately half of adults with ID is estimated to experience communication difficulties. AAC supports them in their daily communication aiming at optimal participation in society. Current communication models, such as Participation Model (Beukelman & Mirenda, 2005) and International Classification of Functioning, Disability and Health (WHO, 2001), regard both client-related and environmental factors as important elements of communication. A substantial part of the environmental factors is made up of the communication partners' characteristics. In daycare and residential services for adults with ID the support worker is an important communication partner .

DETAILED DESCRIPTION:
This study aims to:

1. with regard to teaching Key Word Signing (KWS), a specific form of AAC, to support workers:

   Analyse the relation between training method, support workers' attitude, and short and long term sign knowledge.
2. with regard to the use of manual signs in everyday communication between support workers and adults with ID:

   * Identity the support workers' characteristics that may influence the quality/quantity of the communication between adults with ID who use manual signs and their support worker.
   * Analyse the nature of this influence as well as any possible interaction effects with the clients' characteristics.
3. Assess whether an existing instrument, designed for measuring interactions between parents and children with cerebral palsy using AAC, may be used with adults client and support workers.

ELIGIBILITY:
Inclusion Criteria:

* uses AAC with client
* client has congenital intellectual disability
* supports client for at least 6 months

Exclusion Criteria:

* client has dementia symptoms
* client has severe, non-corrected visual impairment
* client has diagnosed autism

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Support workers who work in residential facilities or day-centres for adults with intellectual disability, in Flanders.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Signing rate of support workers and individuals with intellectual disabilities | Three observation sessions over period of 2 weeks per participant, 2 years for all participants
  Proportion: number of signed utterances divided by total number (spoken + exclusively spoken) of utterances
Sign imitation rate support workers and individuals with intellectual disabilities | Three observation sessions over period of 2 weeks per participant, 2 years for all participants
  Proportion: number of manual sign imitations divided by total number manual signs produced

SECONDARY OUTCOMES:
Explicit Attitude of direct care staff towards manual signs | One testing per participant, over period of 6 months for all participants
  Self-developed survey with subscales (Likert response): scaled score
Implicit Attitude of direct care staff working in towards manual signs | One testing per participant, over period of 6 months for all participants
  Single-Category Implicit Association Test scores
Communicative functions of individuals with intellectual disabilities | Three observation sessions over period of 2 weeks per participant, 2 years for all participants
  Proportion of responses/acknowledgement versus all communicative functions (responses/acknowledgements as well as initiations)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Rombouts, PhD cand., Principal Investigator — KU Leuven
Locations (3):
- Belgium (3):
  - KULeuven, Leuven, Flanders
  - Katholieke Universiteit Leuven, Leuven, Vlaams-Brabant
  - KULeuven, Leuven, Vlaams-Brabant